CLINICAL TRIAL: NCT01235000
Title: TITRE IIB Follow-Up: TIV Infant/Toddler Response Evaluation - Follow-up for Influenza B Boost
Brief Title: TIV Infant/Toddler Response Evaluation - Follow-up for Influenza B Boost
Acronym: TITRE IIB
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: British Columbia Centre for Disease Control (Other Government)
Responsible Party: Dr. Danuta M. Skowronski, BC Centre for Disease Control
Other Study IDs: CIHR 200903CVC-203708/99971a
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Influenza
Keywords: Influenza vaccines; Infant; Dose-Response relationship, immunologic; Prime-boost response
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2010-11 influenza vaccine recipients: Participants of an earlier clinical trial (TITRE II) to evaluate prime-boost response across B lineages in 2009-10
  Interventions: Biological: 2010-11 trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: 2010-11 trivalent inactivated influenza vaccine — A single age-appropriate dose of 2010-11 trivalent inactivated influenza vaccine

SUMMARY:
Each winter, viruses belonging to two kinds of influenza A ("A/H1N1" & "A/H3N2") and two kinds of influenza B ("B/Yamagata" & "B/Victoria") can cause illness. The yearly influenza vaccine is designed to protect against both kinds of influenza A but only one or the other kind of influenza B. Current recommendations in Canada are that if an eligible child less than nine years of age has received two doses of influenza vaccine before, then that child only requires a single dose of influenza vaccine in subsequent years of immunization. In a previous study conducted in early 2010 we measured the antibody response to influenza B in children who had previously received two doses of a B/Yamagata kind of virus contained in the 2008-09 influenza vaccine and just one dose of the B/Victoria kind of virus contained in the 2009-10 recommended vaccine. The purpose of this follow-up study is to see if the protection (antibodies in the blood) provided against the influenza B/Victoria kind of virus that was in the 2009-10 vaccine can be improved with another (second) dose of the same B/Victoria kind of virus included in the 2010-11 vaccine. Since influenza B is an illness especially of children, understanding how to best protect children against both kinds of influenza B is important.

ELIGIBILITY:
Inclusion Criteria:

* Child previously participated in the TITRE II study;
* Child is healthy (stable chronic conditions acceptable) as established by health assessment interview and verbal history-directed health examination;
* Child is available and can complete all relevant procedures during the study period;
* Parent or legal guardian is available and can be reached by phone during the study period;
* Parent/guardian provides written informed consent;
* And, parent/guardian is fluent in English/French.

Exclusion Criteria:

* Child has already received the 2010-11 seasonal (TIV) influenza vaccine
* Child has received immune globulin or other blood products within the prior six weeks;
* Child has received injected or oral steroids within prior six weeks;
* Child is or will be enrolled in any other clinical trial of a drug, vaccine or medical device during the study period;
* Or, child has a recently acquired health condition which, in the opinion of the investigator, would interfere with the evaluation or pose a health risk to the child.

Ages: 29 Months to 51 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants of an earlier clinical trial (TITRE I); enrolled in winter 2008/09 as previously unimmunized infants and toddlers (6-23 months of age) who later participated in 2009-10 study (TITRE II) to receive 2009-10 influenza vaccine
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-10

PRIMARY OUTCOMES:
The seroprotection rate for B/Brisbane/60/2008(Victoria)-like and B/Florida/4/06(Yamagata)-like viruses | 4-6 weeks following a single dose of 2010-11 trivalent inactivated influenza vaccine (TIV)
  The seroprotection rate based on hemagglutination inhibition (HI) assay for B/Brisbane/60/2008(Victoria)-like and B/Florida/4/06(Yamagata)-like viruses following a single age-appropriate dose of 2010-11 TIV containing B/Brisbane/60/2008(Victoria)-like virus in young children originally primed with two doses of 2008-09 TIV containing B/Florida/4/2006(Yamagata) and who had received a single dose of the 2009-10 TIV containing B/Brisbane/60/2008(Victoria) virus

SECONDARY OUTCOMES:
Antibody response to other relevant TIV components | 4-6 weeks following a single dose of 2010-11 TIV
  Other indicators of antibody response to each of the relevant TIV components will also be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Danuta M Skowronski, MD, Principal Investigator — BC Centre for Disease Control, Vancouver, Canada
Locations (3):
- Canada (3):
  - BC Centre for Disease Control, Vancouver, British Columbia
  - McGill University Health Centre - Vaccine Study Centre, Montreal, Quebec
  - Université Laval - Unité de recherche en santé publique, Québec, Quebec

REFERENCES:
- [Derived] Skowronski DM, Hottes TS, De Serres G, Ward BJ, Janjua NZ, Sabaiduc S, Chan T, Petric M. Influenza Beta/Victoria antigen induces strong recall of Beta/Yamagata but lower Beta/Victoria response in children primed with two doses of Beta/Yamagata. Pediatr Infect Dis J. 2011 Oct;30(10):833-9. doi: 10.1097/INF.0b013e31822db4dc. PMID 21857263